CLINICAL TRIAL: NCT06636305
Title: Postpartum Behavioral Observation of Diet, Image, and Exercise Study (BODIES)
Brief Title: Investigation of Increased Physical Activity During the Postpartum Period on Weight Loss, Body Composition, and Energy Expenditure
Acronym: BODIES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolas D. Knuth (Other)
Responsible Party: Sponsor-Investigator, Nicolas D. Knuth, Associate Professor, Towson University
Organization: Towson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1707021250
Record Dates: First submitted 2024-10-04; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Weight Loss; Postpartum; Physical Activity
Keywords: Postpartum; Weight Loss; Physical Activity
MeSH Terms: conditions — Weight Loss; Motor Activity

STUDY DESIGN:
Intervention Model Description: One groups will be assigned to a physical activity intervention, the other group will serve as a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- physical activity intervention (Experimental): Women in the intervention group were instructed to obtain 10,000 steps per day and 150 minutes of MVPA (defined as physical activity that resulted in a heart rate in the range of 120-170 bmp) per week and were given a physical activity tracker (FitBit Charge HR 2, Fitbit, San Francisco, USA) to self-monitor progress.
  Interventions: Behavioral: physical activity intervention
- control group (No Intervention): Women in the control group were given a physical activity tracker (FitBit Charge HR 2, Fitbit, San Francisco, USA) but no other physical activity instructions.

INTERVENTIONS:
Behavioral: physical activity intervention — Women in the intervention group were instructed to obtain 10,000 steps per day and 150 minutes of MVPA (defined as physical activity that resulted in a heart rate in the range of 120-170 bmp) per week and were given a physical activity tracker (FitBit Charge HR 2, Fitbit, San Francisco, USA) to self-monitor progress.
  Arms: physical activity intervention

SUMMARY:
The overall goal of this study is to investigate the impact of increased physical activity during the postpartum period on on weight loss, body composition, energy expenditure, and body image perceptions following pregnancy and childbirth. Specifically, this study utilizes a mixed methods approach including qualitative and quantitative analyses of the physiological and sociological determinants of postpartum women's health and wellness,

The primary objective of the proposed project is to assess the impact of a physical activity intervention on postpartum women's ability to return to pre-pregnancy body weight, the resumption of normal activity and bodily function, and the improvement of body image.

This objective will be achieved via the assessment of quantitative, physiological markers (i.e. physical activity level, body composition, energy expenditure, and hormone levels), as well as qualitative, sociological markers (i.e. self-report and interview data related to body image and bodily recovery) that serve as a measure of a postpartum body that has resumed relatively normal physical function and activity.

DETAILED DESCRIPTION:
Postpartum women will be recruited to participate and randomly assigned to a control group or an intervention group. Both groups will follow the data collection protocol described below; however, the intervention group will also be tasked with a self-administered physical activity intervention while the control group will be told to go about their normal routine and engage in whatever activity they would normally do. The intervention group will be asked to meet physical activity benchmarks of 10,000 steps per day and 150 minutes of moderate-to-vigorous physical activity (MVPA) per week (intervention protocol described in more detail below).

All participants will begin the study when they are between 6 weeks and 3 months postpartum and, overall, data will be collect at 4 separate visits, approximately 3 months apart, over the course of 9 months.

Testing to occur at each visit:

Body composition - Total fat mass, lean tissue mass and percentage of body fat will be assessed as participants lie in a supine position using dual-energy x-ray absorptiometry (DXA) (GE Lunar Prodigy, GE Medical Systems, Milwaukee WI).

Vascular Function Test - Indices of vascular function will be obtained in the non-dominant arm using a strain gauge plethsymograph or ultrasound. The testing entails wrapping a rubber band like device (i.e., strain gauge) around the forearm or placing an ultrasound on the skin while the subject is in a supine position. To induce a change in blood flow, a blood pressure cuff is wrapped around the upper portion of the limb (upper arm or thigh) and occluded for 5 minutes. After the 5 minute occlusion the blood pressure cuff is rapidly deflated. The change in the diameter of the strain gauge is used to quantify the change in blood flow and, in turn, the change in vascular function.

Resting energy expenditure (REE) - REE represents the minimum amount of energy the body needs to maintain normal body function and will be measured while fasted by indirect calorimetry over 20-30 minutes while lying down comfortable.

Blood draw - A 15mL blood draw will be made to allow measurement of metabolic substrate (glucose, fatty acids, triglycerides, cholesterol) and inflammation factors (IL-6, IL-1, TNF-a) related to metabolic rate and fatigue.

Blood pressure, height & weight measurements.

Surveys and monitoring to be administered and/or completed at each visits 1:

Participant Information Form - requires participant to list their name and contact information as well as relevant physician and emergency contact information.

Medical History Form -Measures self-reported general health history. Participants will only complete this form at visit 1.

Pittsburg Sleep Quality Index (PSQI) - a self-rated questionnaire assessment that measures sleep quality and disturbance over a 1-month time interval. Nineteen items generate scores to assess sleep quality, latency and duration.

Demographic Survey - Measures self-reported demographic characteristics of the participants. Participants will only complete this form at visit 1.

Breastfeeding Questionnaire - Asks questions about breastfeeding practices

3-day food record- Allows quantifying and qualifying diet over a 3 day period. Participants will take this form home to complete and return at visits 2, 4, & 6.

Body Image Quality of Life Inventory (BIQLI) - Self-reported 7-point response format ranging from very negative (-3) to very positive (+3) to assess effects of body image on 19 life domains (including sense of self, social functioning, sexuality, emotional well-being, eating, exercise, grooming, etc.).

Edinburg Postpartum Depression Scale (EDPS) - The EDPS is a self-reported 10-item psychological rating scale for measuring the severity of postnatal depression symptoms. This is a standard scale utilized in clinical settings (OBGYN, Pediatrician, & specialized clinician visits).

Multidimensional Assessment of Fatigue (MAF) - This is a self-reported 16-item rating scale useful in measuring the experience of fatigue and its relationship to one's ability to execute daily activities and perform tasks/roles.

Daily activity and sleep monitoring (7 consecutive days)- Objective sleep and physical activity data will be collected using wristwatch actigraph technology. The device is worn on the non-dominant arm and provides accurate and reliable activity and sleep time measurements, including; number of steps taken, estimated energy expenditure, amount of sleep, frequency of awakenings and sleep efficiency. This device has been well validated. Participants will be fitted with this device and wear it for 7 consecutive days.

American College of Obstetricians & Gynecologists (ACOG) Brochure "Exercise after Pregnancy" - This pamphlet explains the benefits of exercise, the latest guidelines for physical activity and details an example of how postpartum women can exercise following pregnancy.

Continuous data collection over nine month period:

Fitbit Data Collection - Participants will be given a Fitbit Charge HR 2 and asked to wear the device for the duration of the study as it will assist them with tracking and achieving step count and MVPA goals. Participants will be asked to consent to share the data the FitBit collects related to daily step count, calories burned, heart rate, and physical activity monitoring. FitBit data will be collected via Fitabase, a research platform that collects data from FitBit devices. The research team will monitor participant FitBit data via Fitabase and send participants assigned to the invertention group weekly text messages regarding their weekly performance. Participants assigned to the control group will not receive weekly feedback regarding their performance.

Specific details of the Intervention Protocol:

The intervention group will be asked to meet physical activity benchmarks of 10,000 steps per day and 150 minutes of MVPA per week (ACOG FAQ Handout entitled "Exercise after pregnancy" will be provided to participants to help define MVPA and provide suggestions for how to engage in physical activity - form attached). MVPA will be defined as physical activity that places heart rate in the range of 120-170 beats per min (bpm) as tracked by the FitBit. Participants will also receive weekly text messages regarding their adherence to the intervention and have access to a brief video that addresses the importance of postpartum physical activity.

ELIGIBILITY:
Inclusion Criteria:

* between 6-12 weeks postpartum following a live singleton birth.

Exclusion Criteria:

* inability to walk without assistance.
* not cleared by their medical provider to resume physical activity by 12 weeks postpartum.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Postpartum Weight Retention | From enrollment to the end of the study at the 12 month postpartum mark
  Postpartum weight retention was calculated as the difference between the participant's postpartum weight at each visit and their self-reported pre-pregnancy weight.

SECONDARY OUTCOMES:
Postpartum Resting Energy Expenditure | REE was measured at enrollment (i.e., 6-12 weeks postpartum) and again at 6, 9, and 12 months postpartum.
  Resting energy expenditure (REE) was measured in supine position for 20 minutes by indirect calorimetry following a >8h fast. REE was calculated from the average rate of oxygen consumption and carbon dioxide production over the last 15 minutes of the test.
Postpartum Body Composition | Postpartum body composition was measured at enrollment (i.e., 6-12 weeks postpartum) and again at 6, 9, and 12 months postpartum.
  Body composition (i.e., fat mass (kg) and fat-free-mass (kg)) was measured by dual energy x-ray absorptiometry. In instances where participants supine body width exceeded the dimensions of the scan window, the analysis of the scans utilized the MirrorImage application.
Postpartum Sleep Quality | Postpartum sleep quality was measured at enrollment (i.e., 6-12 weeks postpartum) and again at 6, 9, and 12 months postpartum.
  The Pittsburg Sleep Quality Index (PSQI) was used to assess sleep quality over the past month at each visit. The PSQI is a 19-item self-report questionnaire indexing seven clinically formulated sleep domains: subjective sleep quality, sleep latency, sleep duration, sleep duration, habitual sleep efficiency, sleep disturbances, and use of sleep medications. Scores on each of the seven PSQI subscales were used to calculate a global score ranging from 0 to 21, with higher score reflecting poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Towson University, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: Access to study IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). Please contact corresponding author for more information or to submit a request.